CLINICAL TRIAL: NCT00951327
Title: Cholangioscopy Using Narrow Band Imaging (NBI) in Patients With Primary Sclerosing Cholangitis (PSC) Undergoing ERCP.
Brief Title: Cholangioscopy Using Narrow Band Imaging (NBI) in Patients With Primary Sclerosing Cholangitis (PSC) Undergoing Endoscopic Retrograde Cholangiopancreatogram (ERCP)
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Todd H. Baron MD, Mayo Clinic
Other Study IDs: 08-006221
Record Dates: First submitted 2009-07-31; First posted 2009-08-04 (Estimated); Last update posted 2010-08-04 (Estimated); Status verified 2010-08

CONDITIONS: Primary Sclerosing Cholangitis
Keywords: Primary sclerosing cholangitis
MeSH Terms: conditions — Cholangitis, Sclerosing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients with primary sclerosing cholangitis (PSC) are affected by an inflammatory condition of the bile ducts. Unfortunately, patients with PSC have a 10 to 15 percent lifetime risk of developing gallbladder and bile duct cancers. Gallbladder and bile duct cancers have a five-year survival of only 5 to 10 percent. Surgery to provide a cure must remove all cancer confined to one area.

In order to increase survival rates there is a need to identify cancer and pre-cancer early. This has been difficult to do.

Patients who have lab tests, positive imaging tests or obstructions will usually have a test called ERCP (Endoscopic Retrograde Cholangiopancreatogram) to take biopsies and enlarge bile ducts or opening bile ducts with stents. Patients usually have cells in the bile ducts removed and analyzed, but there are not studies to show how sensitive this may be to determine if the cells are cancer or pre-cancerous. A new scope with a system using light filters called Narrow Band Imaging (NBI) may help detect cancer and pre-cancer more often and at an earlier stage.

ELIGIBILITY:
Inclusion Criteria:

* Patients with PSC presenting for ERCP where tissue sampling is indicated
* Adults age 18 to 75 years old
* Able to give informed written consent
* Either male or female

Exclusion Criteria:

* PSC with acute cholangitis
* Patients with acute or chronic, debilitating cardiopulmonary disease who are unable to safely undergo prolonged conscious sedation
* Patients with a prior history of liver transplant
* Prisoners
* Unable or unwilling to give informed consents

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting for ERCP with history of Primary Sclerosing Cholangitis
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2008-11; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Cholangioscopy with NBI will enhance the ability to identify sites of potential dysplasia or malignancy in patients with PSC and will be more sensitive in identifying dysplasia than ERCP with biliary brushing and fluoroscopy-guided forceps biopsy. | One year

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Azeem N, Gostout CJ, Knipschield M, Baron TH. Cholangioscopy with narrow-band imaging in patients with primary sclerosing cholangitis undergoing ERCP. Gastrointest Endosc. 2014 May;79(5):773-779.e2. doi: 10.1016/j.gie.2013.09.017. Epub 2013 Oct 24. PMID 24206748